CLINICAL TRIAL: NCT07019233
Title: Effect of Real-time Pressure Controllers on Objective and Subjective Symptoms of Albumin Paclitaxel-induced Peripheral Neuropathy: a Prospective Controlled Research Project
Brief Title: A Study of the Effect of Real-time Pressure Controllers on Subjective and Objective Symptoms of Peripheral Neuropathy Induced by Albumin Paclitaxel
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TJIA2025
Record Dates: First submitted 2025-05-15; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Real Time Pressure Controller; Breast Cancer; Albumin Paclitaxel; Peripheral Neuropathy
MeSH Terms: conditions — Breast Neoplasms; Peripheral Nervous System Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No intervention (No Intervention)
- two-handed intervention (Experimental)
  Interventions: Device: Real Time Pressure Controller

INTERVENTIONS:
Device: Real Time Pressure Controller — The purpose of the real-time pressure controller proposed in this experiment is to overcome the deficiencies of the existing technology and provide a pressure filling device for the prevention of chemotherapy-induced peripheral neuropathy that can accurately control the pressure, with the pressure decreasing in a sequential manner from the distal end (toes/fingers) to the proximal end (wrists, limbs). The application of this device is of great clinical significance to reduce the peripheral neurotoxicity of paclitaxel and to improve patients' drug compliance.
  Arms: two-handed intervention

SUMMARY:
The purpose of the real-time pressure controller proposed in this experiment is to overcome the deficiencies of the existing technology and provide a pressure filling device for the prevention of chemotherapy-induced peripheral neuropathy that can accurately control the pressure, with the pressure decreasing in a sequential manner from the distal end (toes/fingers) to the proximal end (wrists, limbs). The application of this device is of great clinical significance to reduce the peripheral neurotoxicity of paclitaxel and to improve patients' drug compliance. The application of cold compresses or gloves or socks with certain wrapping force is not suitable for the Chinese population, and the acceptance degree of Chinese patients is poor, and the pressure gloves lack individual specificity, and the precise control of pressure for real-time regulation cannot be realized, and the clinical effect is relatively poor. The purpose of this utility model device is to overcome the deficiencies of the existing technology, to provide a pressure filling device for the prevention of chemotherapy-induced peripheral neuropathy that can accurately control the pressure, and the pressure decreases in a sequential manner from the distal end (toes/fingers) to the proximal end (wrist, limb). After applying for the patent, it will be transformed into the market, which has a vast space of medical benefits and market benefits. Paclitaxel is the cornerstone drug in breast cancer chemotherapy, and the neuropathy it causes is often a key factor leading to drug reduction or discontinuation, so opening up the prevention of peripheral neuropathy caused by paclitaxel is of great clinical use.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed written informed consent;
2. Age ≥18 years and ≤75 years at enrollment, male or female patients;
3. Eastern Cooperative Oncology Group (ECOG) physical status score of 0 or 1;
4. Suitable for albumin-paclitaxel antitumor therapy;
5. Cardiopulmonary, hepatic, renal, and coagulation functions are basically normal.

Exclusion Criteria:

1. Patients with prior chemotherapy;
2. Patients with a prior diagnosis of peripheral neuropathy;
3. Patients with a prior diagnosis of associated comorbidities (e.g., diabetes mellitus).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CIPN-related symptoms, as assessed by changes in tactile sensitivity at pretreatment baseline CIPN incidence.The Patient Neurotoxicity Questionnaire (PNQ) was used to assess and grade the incidence and severity of CIPN. | through study completion, an average of 1 year
  From the time a patient begins albumin paclitaxel therapy until the patient's treatment on this regimen is completed, or during albumin paclitaxel therapy, adverse reactions due to pressure gloves that result in patient patient disenrollment or voluntary.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, China

IPD SHARING:
Plan to Share IPD: No